CLINICAL TRIAL: NCT02833103
Title: Application of Pinaverium Bromide in the Treatment of Patients With Post-cholecystectomy Sphincter of Oddi Dysfunction (SOD): A Randomized, Controlled and Multicenter Clinical Study
Brief Title: Pinaverium Bromide in Post-cholecystectomy Sphincter of Oddi Dysfunction
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Zhaohui Tang, the chief surgeon of the department of General Surgery, Xinhua Hospital, Shanghai Jiao Tong University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: XH-16-015
Record Dates: First submitted 2016-07-04; First posted 2016-07-14 (Estimated); Last update posted 2016-07-14 (Estimated); Status verified 2016-07

CONDITIONS: Sphincter of Oddi Dysfunction
Keywords: Pinaverium Bromide; cholecystectomy; Sphincter of Oddi Dysfunction
MeSH Terms: conditions — Sphincter of Oddi Dysfunction | interventions — pinaverium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pinaverium Bromide group (Experimental): Able to improve the spasms of SO; literature showed that it treated biliary disorders effectively.
  Interventions: Drug: Pinaverium Bromide
- Danshu group (Active Comparator): Contains the active pharmaceutical ingredient (API) and has the effects of fighting infection, alleviating pain, promoting bile secretion and lifting muscle spasms; literature showed that Danshu Capsules effectively improved the symptoms of biliary disorders, such as pain, nausea and abdominal distension.
  Interventions: Drug: Danshu Capsules

INTERVENTIONS:
Drug: Danshu Capsules — Danshu Capsules (0.9g potid/day) for three months by oral
  Other Names: Danshu softgel Capsules
  Arms: Danshu group
Drug: Pinaverium Bromide — Pinaverium Bromide (100mg potid/day) for three months by oral
  Other Names: Dicetel
  Arms: Pinaverium Bromide group

SUMMARY:
Sphincter of Oddi dysfunction (SOD) refers to biliary kinetic abnormality of the sphincter of Oddi (SO), often accompanied by pain, hepatic and pancreatic enzyme elevation, common bile duct (CBD) dilation or onset of pancreatitis. Pain caused by SOD affects the quality of life (QoL).The primary objective of this trial is to evaluate the efficacy of relieving abdominal pain of Pinaverium Bromide in medication therapy for patients with post-cholecystectomy SOD.

DETAILED DESCRIPTION:
1.1 Background (I)

1.1.1 10%~50% of the patients who previously underwent cholecystectomy experience recurrent abdominal pain with or without diarrhea, abdominal distention, enzymatic changes, etc., and sphincter of Oddi dysfunction (SOD) accounts for about 13% of such cases;

1.1.2 Sphincter of Oddi dysfunction (SOD):

* It refers to biliary kinetic abnormality of the sphincter of Oddi (SO), often accompanied by pain, hepatic and pancreatic enzyme elevation, common bile duct (CBD) dilation or onset of pancreatitis.
* Pain caused by SOD affects the quality of life (QoL).

1.1.3 The diagnosis of SOD is still being disputed, and there has been no optimal solution so far.

* The diagnosis of SOD is largely based on clinical judgment
* The gold standards ERCP and SOM are invasive diagnostic criteria

1.2 Background (II)

1.2.1 If biliary-type abdominal pain after cholecystectomy is considered as SOD, most of the patients are classified as SOD II and SOD III according to Rome III Criteria-modified.

Biliary SOD Type I: moderate or severe biliary-type abdominal pain; transient ALT / AST/ALP elevation > 2ULN; CBD dilation > 8mm as evidenced by ultrasound or other non-invasive examination Type II: biliary-type abdominal pain; One or two of above items Type III:only biliary-type abdominal pain

1.3 Background (III)

1.3.1 Treatment of SOD is being disputed: currently, the main method is to relax sphincter of Oddi (SO).

* Medications: antispasmodic drugs, nitrates, calcium ion antagonists, modulators of gastrointestinal (GI) motility
* EST(endoscopic sphincterotomy): postoperative complications and mortality

1.3.2 EST is not well effective in the treatment of SOD type II and type III, which are mostly caused by functional abnormalities

-ASGE guideline 2015 points out that EST is not recommended for patients with SOD type III. Endoscopic stents are not recommended, either.

1.3.3 Danshu Capsules: contains the active pharmaceutical ingredient (API) and has the effects of fighting infection, alleviating pain, promoting bile secretion and lifting muscle spasms; literature showed that Danshu Capsules effectively improved the symptoms of biliary disorders, such as pain, nausea and abdominal distension.

1.3.4 Pinaverium Bromide: able to improve the spasms of SO; literature showed that it treated biliary disorders effectively.·10%~50% of the patients who previously underwent cholecystectomy experience recurrent abdominal pain with or without diarrhea, abdominal distention, enzymatic changes, etc., and sphincter of Oddi dysfunction (SOD) accounts for about 13% of such cases.

ELIGIBILITY:
Inclusion Criteria:

* Chief complaint of upper right abdominal pain following LC (within 2 weeks to 6 months) at a hospital visit, but not a pain caused by surgical incision, lasting 3 to 5 minutes each time, without a history of other biliary tract operation
* No presence of intestinal obstruction as evidenced by plain abdominal X-ray, with peptic ulcer and duodenal diverticulum ruled out through barium meal examination or gastroscopy
* No other obvious abnormalities as evidenced by abdominal ultrasound B and MRCP, except for bile duct dilation
* Patients with biliary-type sphincter of Oddi dysfunction (SOD) who are classified as SOD type II (biliary-type abdominal pain accompanied by hepatic enzyme elevation or common bile duct (CBD) dilation) and SOD type III (only biliary-type abdominal pain) according to Geenen-Hogan classification criteria

Exclusion Criteria:

* Postoperative biliary calculi, benign biliary stenosis, bile duct infection, overlong residual cystic duct (> 0.5cm), biliary tumors, etc.
* Peptic ulcer, duodenal diverticulum
* Pancreatitis, pancreatic-type SOD
* Adhesive intestinal obstruction
* Postoperative irritable bowel syndrome (IBS)
* A history of abdominal operation or other surgery
* Pregnant and lactating women
* Use of other drugs from one week after LC to enrollment, including antispasmodic drugs, analgesics, choleretic agents, calcium ion antagonists and GI motility drugs
* A history of allergy to Pinaverium Bromide / Danshu Tablets

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Estimated)
Dates: Start 2016-07; Primary Completion 2018-02 (Estimated); Study Completion 2018-02 (Estimated)

PRIMARY OUTCOMES:
Efficacy Evaluation of Reduction in Abdominal Pain Scores，Change From Baseline to 3 Months After Medication | Change From Baseline to 3 Months After Medication
  abdominal pain scores (baseline vs. 3 months after treatment)
  * Abdominal pain score based on main symptom: Degree of pain in point（0 - no pain [0 point]；1~3 - mild pain [1 point]；4~6 moderate pain [2 point]]；7~10 - severe pain [3 point]）、Frequency in times/week (No episodes[0 point]；1 time/week[1 point]；2 times/week[2 point]; 3 times/week[3 point])、Duration in days/week(No episodes[0 point]；< 1 day/week[1 point]；1-2days/week[2 points]；≥ 3days/week[3 points])
  * The sum of the scores for the above three items is the total score for abdominal pain.
  * Efficacy evaluation: reduction in abdominal pain score, as compared with the baseline
  * = 100%: complete remission (CR)；60%~99%: significant remission (SR)；30% ~ 59%: partial remission (PR)；0% ~ 29%: no response (NR)
  * Treatment response = CR + SR
  * Treatment response rate = (CR + SR) / the total number of patients

SECONDARY OUTCOMES:
Changes in the Common Bile Duct (CBD) Diameter Measured by Ultrasound B Once a Month | Once a Month, Four Times Totally (baseline / 4w after treatment / 8w after treatment / 12w after treatment)
  Changes in the CBD diameter measured by ultrasound B
  * Each patient is required to abstain from eating for 12 hours and then takes a measurement of the CBD diameter by ultrasound B the next morning
  * The measurement takes places once a month, four times totally (baseline / 4w after treatment / 8w after treatment / 12w after treatment)
Efficacy of Lowering Liver Enzymes as Assessed by Laboratory Test Once a Month | Once a Month, Four Times Totally (baseline / 4w after treatment / 8w after treatment / 12w after treatment)
  * Changes in hepatic enzyme levels (ALT, AST and ALP)
  * The measurement takes place once a month, four times totally (baseline / 4w after treatment / 8w after treatment / 12w after treatment)
Number of Participants With Treatment-Related Diarrhea,Change From Baseline to 3 Months After Medication | From Baseline to 3 Months After Medication
  The number of patients presenting the symptoms of diarrhea will be calculated at the time of enrollment (baseline) and 3 months after treatment respectively.

OTHER OUTCOMES:
Number of Participants With Treatment-Related Adverse Events as Assessed by Researchers or Doctors Through Study Completion | Through Study Completion, An Average of 1 Year
  Incidence of adverse events (throughout the treatment)
  * The type and number of adverse events will be calculated at the baseline and each visit
  * Inquire about symptoms: rashes, pruritus, acid regurgitation, abdominal distention, diarrhea, etc.
  * Perform the following examinations at the last visit: blood / urine / stool test, liver / kidney function test, ECG

CONTACTS AND LOCATIONS:
Overall Officials: Zhaohui Tang, MD,PhD, Principal Investigator — Xinhua Hospital,School of Medicine,Shanghai Jiao Tong University; Zhiwei Quan, MD,PhD, Study Chair — Xinhua Hospital,School of Medicine,Shanghai Jiao Tong University
Locations (1):
- Zhang Yong, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cotton PB, Durkalski V, Romagnuolo J, Pauls Q, Fogel E, Tarnasky P, Aliperti G, Freeman M, Kozarek R, Jamidar P, Wilcox M, Serrano J, Brawman-Mintzer O, Elta G, Mauldin P, Thornhill A, Hawes R, Wood-Williams A, Orrell K, Drossman D, Robuck P. Effect of endoscopic sphincterotomy for suspected sphincter of Oddi dysfunction on pain-related disability following cholecystectomy: the EPISOD randomized clinical trial. JAMA. 2014 May;311(20):2101-9. doi: 10.1001/jama.2014.5220. PMID 24867013
- [Background] Vitton V, Ezzedine S, Gonzalez JM, Gasmi M, Grimaud JC, Barthet M. Medical treatment for sphincter of oddi dysfunction: can it replace endoscopic sphincterotomy? World J Gastroenterol. 2012 Apr 14;18(14):1610-5. doi: 10.3748/wjg.v18.i14.1610. PMID 22529689
- [Background] Okoro N, Patel A, Goldstein M, Narahari N, Cai Q. Ursodeoxycholic acid treatment for patients with postcholecystectomy pain and bile microlithiasis. Gastrointest Endosc. 2008 Jul;68(1):69-74. doi: 10.1016/j.gie.2007.09.046. PMID 18577477
- [Background] Kalaitzakis E, Ambrose T, Phillips-Hughes J, Collier J, Chapman RW. Management of patients with biliary sphincter of Oddi disorder without sphincter of Oddi manometry. BMC Gastroenterol. 2010 Oct 22;10:124. doi: 10.1186/1471-230X-10-124. PMID 20969779
- [Background] Behar J, Corazziari E, Guelrud M, Hogan W, Sherman S, Toouli J. Functional gallbladder and sphincter of oddi disorders. Gastroenterology. 2006 Apr;130(5):1498-509. doi: 10.1053/j.gastro.2005.11.063. PMID 16678563
- [Background] Drossman DA. The functional gastrointestinal disorders and the Rome III process. Gastroenterology. 2006 Apr;130(5):1377-90. doi: 10.1053/j.gastro.2006.03.008. No abstract available. PMID 16678553
- [Background] Hernando N, Gisler SM, Reining SC, Deliot N, Capuano P, Biber J, Murer H. NaPi-IIa interacting proteins and regulation of renal reabsorption of phosphate. Urol Res. 2010 Aug;38(4):271-6. doi: 10.1007/s00240-010-0304-3. Epub 2010 Jul 28. PMID 20665015